CLINICAL TRIAL: NCT02312986
Title: Use of Fecal Microbiota Transplantation (FMT) to Reverse Multi-Drug Resistant Organism Carriage
Brief Title: FMT for Multidrug Resistant Organism Reversal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201506131
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Infection With Multi-drug Resistant Organisms
Keywords: infection; colonization; antibiotic resistance
MeSH Terms: conditions — Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal microbiota transplantation (Experimental): Subjects will receive 150mL of fecal microbiota product via enema.
  Interventions: Biological: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Biological: Fecal microbiota transplantation (FMT) — Prospective pilot study to examine whether fecal microbiota transplantation (FMT) is able to suppress or reverse gastrointestinal carriage of multi-drug resistant organisms.
  Other Names: FMT; stool transplant

SUMMARY:
This proposed protocol involves the use of the fecal microbiota transplantation (FMT) to suppress or reverse colonization with multidrug resistant organisms (MDRO) in subjects with recurrent MDRO infections due to organisms of likely enteric origin.

FMT will be performed on subjects with a history of at least three recurrent infections due to MDRO; at least two recurrent, severe infections due to MDRO requiring hospitalization; or at least two recurrent infections due to MDRO for which only antimicrobials with rate limiting toxicities are available.

The objective of this protocol is to determine if fecal microbiota transplantation (FMT) will be able to prevent additional recurrences of infections due to MDRO by suppressing or reversing enteric colonization with MDRO.

DETAILED DESCRIPTION:
This is a prospective pilot study of fecal microbiota transplantation in patients with a history of recurrent MDRO infections. Subjects who meet inclusion/exclusion criteria and provide written, informed consent will provide a pre-FMT stool sample. The FMT will be administered by enema in the outpatient setting by trained personnel. Patients will provide stool samples 30 days, 6 months, and 12 months post-FMT. The subjects will also be monitored for potential adverse events, recurrence of MDRO infections, infections that may be related to FMT, and worsening of existing comorbidities or development of new comorbidities.

ELIGIBILITY:
Inclusion criteria will include:

* Age ≥18 years old.
* Outpatient status at time of FMT.
* History of at least three recurrent infections due to an MDRO; at least two recurrent, severe infections due to MDRO requiring hospitalization; or at least two recurrent infections due to MDRO for which only antimicrobials with rate limiting toxicities (see above) are available AND the MDRO is likely of enteric origin. Only MDROs of likely enteric origin will be included.
* Be without active infection due to the MDRO at the time of FMT.
* Not be receiving antimicrobials (therapeutic or suppressive) within 48 hours of FMT.

Exclusion criteria will include:

* Subjects <18 years old.
* Subjects unable to be seen as an outpatient.
* Use of enteral or systemic antimicrobials at time of FMT.
* Planned use of enteral or systemic antimicrobials up to 6 months post-FMT.
* Pregnancy or inability/unwillingness to use contraceptives.
* Recent intra-abdominal surgery
* Short gut syndrome
* Gastrointestinal motility disorders
* Use of medications that affect intestinal motility an inability to cease using those medications at the time of FMT.
* Post-allogeneic hematopoietic stem cell transplant recipients with previous or current gastrointestinal graft versus host disease.
* ANC <500/mm3
* HIV+ and not well controlled on antiretroviral therapy, or CD4+ <200/ mm3
* At increased risk for peritonitis: presence of intra-abdominal devices, receiving peritoneal dialysis, or ascites.
* Any acute illness
* Recurrent C. difficile infection.
* Unlikely to survive for 3 months.
* Investigator feels the risks of FMT outweigh potential benefit, including other conditions or medications that the investigator determines puts the subject at greater risk from FMT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik R Dubberke, MD, MSPH, Principal Investigator — Washington University School of Medicine

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fecal Microbiota Transplantation
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One participant was enrolled in this trial.
Arm/Group | Fecal Microbiota Transplantation
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of FMT in Patients With Recurrent MDRO Infections (Incidence and Severity of Solicited and Serious Adverse Events)
Description: Incidence and severity of solicited and serious adverse events within 12 months of FMT.
Time Frame: 12 months post-FMT
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplantation
Number analyzed (Participants) | 1
Participants
  Solicited adverse events related to FMT | 0
  Any serious adverse event | 1

2. Secondary Outcome: MDRO Infection Status Post-FMT (Number of Subjects With MDRO Infections)
Description: Number of subjects with MDRO infections 30 days, 6 months, and 12 months post-FMT.
Time Frame: 30 days, 6 months, and 12 months post-FMT
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplantation
Number analyzed (Participants) | 1
Participants
  MDRO infection at 30 days | 0
  MDRO infection at 6 months post-FMT | 1
  MDRO infection at 12 months | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Fecal Microbiota Transplantation
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplantation (N=1)
Gangrene (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Oropharyngeal squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fecal Microbiota Transplantation (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02312986/Prot_SAP_000.pdf